CLINICAL TRIAL: NCT04445545
Title: Effectiveness of High Intensity Laser Therapy (HILT) and Stretching Exercises on Cervical Flexibility and Pain Reduction in Myofascial Trigger Points. Randomized Clinical Trial (RCT).
Brief Title: High Intensity Laser Therapy (HILT) on Myofascial Trigger Points.
Acronym: HILT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 60312070
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Myofascial Trigger Point Pain (MTrP)
Keywords: Lasers; Laser Therapy; Trigger Points; Myofascial Pain Syndromes; Analgesia; Clinical Trial
MeSH Terms: conditions — Myofascial Pain Syndromes; Agnosia | interventions — Ultrasonic Therapy; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (HILT + stretching exercise) (Experimental): The group will receive treatment of high-intensity laser therapy (HILT) with a total energy delivery of 1,060J divided into 3 phases will be achieved: phase 1, 500J; phase 2, 60J; phase 3, 500J. It will work with an average power of 3W and an energy density of 50J/cm2. At the end of the assigned treatment will be added a treatment protocol of upper trapezius stretching exercises for the evaluated limb with shortening. The stretches will consist of 4 series of 30 seconds with an interval of 30 seconds between series.
  Interventions: Device: High intensity laser therapy (HILT); Procedure: Stretching exercise
- Experimental group 2 (Sham HILT + stretching exercise) (Sham Comparator): The group will receive a sham treatment of high-intensity laser therapy (HILT). At the end of the assigned treatment will be added a treatment protocol of upper trapezius stretching exercises for the evaluated limb with shortening. The stretches will consist of 4 series of 30 seconds with an interval of 30 seconds between series.
  Interventions: Device: High intensity laser therapy (HILT); Procedure: Stretching exercise
- Experimental group 3 (US + stretching exercise) (Active Comparator): The group will receive treatment of therapeutic ultrasound. The US parameters will be programmed with a frequency of 1MHz, the intensity of 1.5 W/cm2, the Duty cycle of 100%, an ERA of 5cm2, and a time of 6 minutes. At the end of the assigned treatment will be added a treatment protocol of upper trapezius stretching exercises for the evaluated limb with shortening. The stretches will consist of 4 series of 30 seconds with an interval of 30 seconds between series.
  Interventions: Device: Therapeutic Ultrasound (US); Procedure: Stretching exercise

INTERVENTIONS:
Device: High intensity laser therapy (HILT) — Laser application with powers greater than 500 milliwatts (mW) in the myofascial trigger point and muscle belly of the upper trapezius. Laser therapy will be applied to the upper trapezius muscle with a total energy delivery of 1,060J divided into 3 phases will be achieved (phase 1, 500J; phase 2, 60J; phase 3, 500J). It will work with an average power of 3W and an energy density of 50J/cm2. For the application of laser therapy, the 12W BTL-6000 equipment that emits infrared wavelengths of 1064nm will be used.
  Arms: Experimental group 1 (HILT + stretching exercise); Experimental group 2 (Sham HILT + stretching exercise)
Device: Therapeutic Ultrasound (US) — Application of ultrasound therapy in the myofascial trigger point of the upper trapezius muscle. The ultrasound application will be performed with the person in a seated position. The ultrasound parameters will consist of a frequency of 1MHz, the intensity of 1.5 W/cm2, a Duty cycle of 100%, an ERA of 5cm2, and a treatment time of 6 minutes.
  Arms: Experimental group 3 (US + stretching exercise)
Procedure: Stretching exercise — t the end of the assigned treatment will be added a treatment protocol of upper trapezius stretching exercises for the evaluated limb with shortening. The stretches will consist of 4 series of 30 seconds with an interval of 30 seconds between series

SUMMARY:
The aim of the study is to evaluate the effects of HILT on cervical flexibility and pain reduction in myofascial trigger points. The research will be carried out in the Physiotherapy laboratory of Andrés Bello University. The participants will be civil servants and volunteer university students with the presence of latent MTrPs of the upper trapezius muscle. Participants will be randomized and divided into 3 study groups: group 1 (HILT and stretching exercises), group 2 (sham HILT and stretching exercises), and group 3 (the conventional US and stretching exercises). The treatments will be carried out twice a week for 4 weeks accompanied by 2 evaluations during the treatment and 1 post-treatment follow-up. The main result will be considered the differences in pain intensity (ΔPI), pain pressure threshold (ΔPPT), cervical spine range (ΔCROM), and cervical disability (ΔND) between the evaluation sessions.

DETAILED DESCRIPTION:
Material and Methods

Type of study: Experimental, randomized clinical trial (RCT).

1. Study population.

For the study, students and workers of Andrés Bello University will be considered participants.

2 Randomization and sample.

Participants will be evaluated according to the selection criteria through a survey with closed questions and a clinical examination in which the presence or absence of shortening of upper trapezius muscle shortening will be determined and the presence of a myofascial trigger point (MTrPs) in the muscle. The participants will be chosen according to the selection criteria through a survey with closed questions and a clinical examination in which the presence of muscle shortening of the upper trapezius and the presence of myofascial trigger point in the said muscle. Participants will be divided into three study groups through a simple randomization process; group 1 (HILT), group 2 (sham HILT), and group 3 (HILT). the conventional US). All groups will receive as a basic treatment a therapeutic exercise plan of active static stretching of the upper trapezius muscle of 4 series for 30 seconds. Participants will be scheduled twice a week for four weeks to carry out the assigned treatment.

The sample size will be determined with the G-Power program using a power of 0.85 (1-β), reliability of 95%, an error of 5% (α), and an effect size of d=0.75 (d-Cohen) taking as reference previous studies that have determined the differences in the PPT mean in MTrPs between experimental groups and controls after treatment with HILT.35,49 Based on the above, the sample size is 24 subjects with 8 subjects per group.

3. Procedures

Participants in each group will be evaluated by two independent examiners to determine cervical spine flexibility (CFROM) and pain intensity (PI), considered the main outcome measures of the study. The range of motion will be measured through goniometry, and pain intensity will be evaluated through algometry, establishing the painful pressure threshold (PPT). The PPT values will be evaluated in kg/cm2, while the CFROM will be evaluated in degrees. The PI and CFROM values will be tabulated in an Excel® spreadsheet for each evaluator.

The evaluations will be carried out during the study in 3 instances (T0-T2) including later 1 follow-up evaluation (T3): pretreatment (T0: baseline), second week (T1: 4th session), fourth week (T2: 8th session). ) and fifth week (T3: follow-up). The participants will be summoned twice a week to carry out their corresponding treatments. On the other hand, cervical disability will be evaluated using the cervical disability index (NDI), obtaining the percentage of disability for each of the evaluation instances. On the other hand, the NDI will be applied as a self-report before and after the treatment sessions (T0 and T2).

Once the study is over, the differences in cervical range of motion (ΔCFROM), pain pressure threshold (ΔPPT), pain intensity (ΔPI), and cervical disability (ΔNDI) between the evaluation sessions will be evaluated.

4. Variables

4.1 Conceptual definition of the variables.

* Cervical flexibility (CFROM): physical capacity responsible for the voluntary execution of the maximum joint movement of the cervical spine. The CFROM examination will be performed by the participant in a seated position keeping their back straight and supported by a backrest.
* Pain intensity (PI): magnitude of pain reported by the participants after performing the myofascial trigger point (MTrP) algometry test in the shortened upper trapezius muscle after performing the test. The test of the PI will be performed by the participant in a seated position keeping their back straight and supported by a backrest.
* Painful pressure threshold (PPT): magnitude of pressure referred to as painful by the participant when performing the algometry test on the myofascial trigger point (MTrP) of the shortened upper trapezius muscle. The PPT exam will be performed by the participant in a seated position keeping their back straight and supported by a backrest.
* Cervical disability (ND): level of cervical condition reported by the participants that compromise or may compromise the normal development of their activities of daily living.
* High-Intensity Laser Therapy (HILT): laser application with powers greater than 500 milliwatts (mW) in the myofascial trigger point and muscle belly of the upper trapezius.
* Conventional ultrasound (US): application of ultrasound therapy in the myofascial trigger point of the upper trapezius muscle.
* Stretching exercise (SE): active static stretching for the upper trapezius muscle with the presence of myofascial trigger points (positive MTrPs).26,40,41

4.2 Operational definition of variables.

* Cervical flexibility (CFROM): The maximum cervical ranges of motion (CFROM) will be evaluated through an inclinometer (CROM device), recording the degrees of movement for the coronal, sagittal and horizontal planes (Inter-rater reliability: Extension ICC = 0.98 ( 95% CI 0.95, 0.99); Flexion ICC = 0.89 (95% CI 0.73, 0.96); Left Rotation ICC = 0.95 (95% CI 0.87, 0.98); Right Rotation ICC = 0.92 (95% CI 0.80, 0.97); Tilt left ICC = 0.97 (95% CI 0.91, 0.99), right slope ICC = 0.97 (95% CI 0.93, 0.99).
* Painful pressure threshold (PPT): the painful pressure threshold (PPT) will be quantified by algometry, recording the pressure values in kg/cm2 that generate pain in the MTrPs of the upper trapezius muscle (intra-rater reliability: ICC = 0.92-0.98 (CI not reported; inter-rater reliability: ICC = 0.92 (95% CI 0.85,0.97).) The Baseline® brand pressure algometer will be used for the evaluation.
* Cervical Disability (ND): Cervical disability will be evaluated through the Cervical Disability Index (NDI), an instrument that consists of 10 sections with questions related to symptoms and activities of daily living in which the cervical region is involved. Each section costs questions scored from 0-5, with greater disability being linked to a higher score (inter-rater reliability: ICC = 0.93 (95% CI 0.86, 0.97)).
* High-Intensity Laser Therapy (HILT): High-intensity laser therapy (HILT) will be applied to the upper trapezius muscle using the protocol of the study by Dundar et al.48 A total energy delivery of 1,060J divided into 3 phases will be achieved. (phase 1, 500J; phase 2, 60J; phase 3, 500J). It will work with an average power of 3W and an energy density of 50J/cm2. For the application of laser therapy, the 12W BTL-6000 equipment will be used, which emits infrared wavelengths of 1064nm (ANNEX 7).
* Conventional ultrasound (US): the application of ultrasound will be performed with the person in a seated position. The ultrasound parameters will consist of a frequency of 1MHz, the intensity of 1.5 W/cm2, a Duty cycle of 100%, an ERA of 5cm2, and a treatment time of 6 minutes.32 The application of US will be carried out using the COMBI 500 equipment of the company GYMNA®.
* Stretching exercise (SE): 4 sets of active static stretching of the upper trapezius muscle will be performed. Each series will last 30 seconds followed by a rest interval of 30 seconds.

4.3 Variable type definition

* Cervical flexibility (CFROM): dependent, quantitative, discrete variable.
* Pain intensity (PI): dependent, quantitative, discrete variable.
* Painful pressure threshold (PPT): dependent, quantitative, discrete variable.
* Cervical disability (ND): dependent variable, quantitative, continuous.
* High-Intensity Laser Therapy (HILT): independent, quantitative, continuous variable.
* Conventional ultrasound (US): independent, quantitative, continuous variable.
* Stretching exercise (EE): independent, quantitative, discrete variable.

  5. Study phases

Three phases have been designated for the investigation; 1. Sampling phase, 2. Evaluation phase and 3. Intervention phase.

The sampling phase will consist of the application of the selection survey to all students and officials interested in participating in the study. The survey will be applied to them through the Google Drive® system. All those who meet the selection criteria will be invited to participate in the research. This stage will last two weeks.

The evaluation phase will determine a second filter of the population and will include the participants selected by the selection survey who expressed their consent in writing. At this stage, a clinical examination will be performed to determine the presence of shortening of the upper trapezius muscle and myofascial trigger points. The evaluation of the length of the upper trapezius will be carried out by means of an evaluation of the cervical tilt range, while the assessment of the MTrPs will be carried out next in the upper trapezius muscle using the criteria established in the study by Delphi et al. (expert agreement for the diagnosis of MTrPs), in which at least two of the following criteria must be present: 1. taut band, 2. hypersensitive point and 3. pain referred to the compression of the point.24,25 It will be considered as shortened upper trapezius, that muscle contralateral to the lowest degree of cervical inclination measured with an inclinometer. In the event that both trapezius muscles present the same value in degrees, the one that the participant refers to with greater tension will be considered as shortening. The MTrPs examination will be performed by drawing a line between the spinous process of C7 and the midpoint of the upper border of the ipsilateral acromion next to the trapezius evaluated as short, palpating from medial to lateral in search of a point that meets the criteria. exposed. In cases where more than 1 MTrP was located along the reference line, the most sensitive or painful point will be used as a reference. Participants with a negative (-) physical examination, that is, without the presence of MTrPs in the trapezius muscle shortened according to the protocol will be excluded, while those with a positive physical examination (+) will be able to participate in the study. The evaluation of muscle shortening and the presence of MTrPs will be carried out by a blind evaluator, who will record the laterality of the shortened muscle and the location distance of the MTrPs in a Microsoft Excel® spreadsheet, taking the spinous process of C7 as a reference.

The intervention phase will consist of 8 treatment sessions. The sample will be randomized into three study groups; group 1 (HILT + stretching exercises), group 2 (sham HILT + stretching exercises), and group 3 (conventional US + stretching exercises). All groups will receive as a basic treatment a therapeutic exercise plan of active static stretching of the upper trapezius muscle of 4 series for 30 seconds. The randomization of the sample will be carried out by the director of the study using the simple random sampling process through the research randomizer program (https://www.randomizer.org/). The results of the randomization will only be known by the director of the studio. Demographic variables for each group, including age, sex, and body mass index (BMI), will be tabulated in a Microsoft Excel® program spreadsheet.

Participants in each group will be evaluated by two independent examiners to determine cervical spine flexibility (CFROM) and pain intensity (PI), considered the main outcome measures of the study. The range of motion will be measured through goniometry, and the intensity of pain will be evaluated through algometry, establishing the painful pressure threshold (PPT). The PPT values will be evaluated in kg/cm2, while the CFROM will be evaluated in degrees. The PI and CFROM values will be tabulated in an Excel® spreadsheet for each evaluator.

6. Statistic analysis

The descriptive statistics for the primary variables ΔCFROM, ΔPPT, and ΔNDI will use as analysis measures, means, and standard deviation (x, SD), or median and interquartile range (med, IQR) according to the normality analysis of the data. For secondary variables such as gender, body mass index (BMI), frequencies, and means or medians will be used, respectively, according to the normality analysis of the data.

For the inferential statistical analysis, the Shapiro Wilk (S-Wilk) normality test will be used to determine the distribution of the primary variables, and according to the results, parametric or non-parametric tests will be selected; One-way ANOVA if data are normally distributed or Kruskal Wallis test if variables are not normally distributed. For the statistical analysis, the STATA.v16 program will be used. Once the statistical analysis is done, a month will be considered for the review of the results, approach to the discussion, and conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years of age.
* Officials and students of the Casona las Condes Campus of the Andrés Bello University.
* Presence of myofascial trigger points in the shortened upper trapezius muscle evaluated (expert consensus establishing criteria for the diagnosis of MTrPs, Delphi study).25

Exclusion Criteria:

* Musculoskeletal problems or pathologies of the neck or shoulders in the last 3 months (fractures, sprains, tendinopathies, dislocations, or muscle tears).
* Presence of osteosynthesis materials near shoulders, neck, or surrounding areas.
* Presence of wounds or skin changes in the shoulder and/or neck region (such as psoriasis, scars, or burns).
* Use of analgesic, anti-inflammatory, or muscle relaxant medications for permanent use.
* Neurological changes such as paresthesia, loss of sensitivity (partial or complete), decreased strength, and color changes in the neck, arms, forearms, or hands.
* Diagnosed photosensitivity.
* Presence of solar urticaria or adverse reactions to sunlight.
* Presence of the following conditions: dermatomyositis, systemic lupus erythematosus, hepatic porphyria, cutaneous carcinoid syndrome or pellagra
* Cancer or tumors of any type diagnosed.
* Epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain pressure thereshold (PPT) | Change from Baseline pain pressure thereshold at eight treatment sessions.
  Comparing pain pressure threshold differences on trigger point of trapezius muscle for pre and post-treatment protocol.
Joint Range changes (CFROM) | Change from Baseline joint range changes at eight treatment sessions.
  Comparing maximum cervical range differences for pre and post for pre and post-treatment protocol.

SECONDARY OUTCOMES:
Neck disability | Change from Baseline meck disability at eight treatment sessions.
  Comparing neck disability for pre and post treatment protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Hernán A de la Barra Ortiz, Mg, Principal Investigator — Universidad Andrés Bello
Locations (2):
- Chile (2):
  - Universidad Andrés Bello, Santiago, Las Condes
  - Universidad Andrés Bello, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotler HB, Chow RT, Hamblin MR, Carroll J. The Use of Low Level Laser Therapy (LLLT) For Musculoskeletal Pain. MOJ Orthop Rheumatol. 2015;2(5):00068. doi: 10.15406/mojor.2015.02.00068. Epub 2015 Jun 9. PMID 26858986
- [Background] Hadis MA, Zainal SA, Holder MJ, Carroll JD, Cooper PR, Milward MR, Palin WM. The dark art of light measurement: accurate radiometry for low-level light therapy. Lasers Med Sci. 2016 May;31(4):789-809. doi: 10.1007/s10103-016-1914-y. Epub 2016 Mar 10. PMID 26964800
- [Background] Peplow PV, Chung TY, Baxter GD. Laser photobiomodulation of proliferation of cells in culture: a review of human and animal studies. Photomed Laser Surg. 2010 Aug;28 Suppl 1:S3-40. doi: 10.1089/pho.2010.2771. PMID 20666617
- [Background] Khalkhal E, Razzaghi M, Rostami-Nejad M, Rezaei-Tavirani M, Heidari Beigvand H, Rezaei Tavirani M. Evaluation of Laser Effects on the Human Body After Laser Therapy. J Lasers Med Sci. 2020 Winter;11(1):91-97. doi: 10.15171/jlms.2020.15. Epub 2020 Jan 18. PMID 32099633
- [Background] Vreman HJ, Wong RJ, Stevenson DK. Phototherapy: current methods and future directions. Semin Perinatol. 2004 Oct;28(5):326-33. doi: 10.1053/j.semperi.2004.09.003. PMID 15686263
- [Background] Calderhead RG, Vasily DB. Low Level Light Therapy with Light-Emitting Diodes for the Aging Face. Clin Plast Surg. 2016 Jul;43(3):541-50. doi: 10.1016/j.cps.2016.03.011. Epub 2016 May 6. PMID 27363768
- [Background] Ohshiro T, Ohshiro T, Sasaki K, Kishi K. Picosecond pulse duration laser treatment for dermal melanocytosis in Asians : A retrospective review. Laser Ther. 2016 Jun 29;25(2):99-104. doi: 10.5978/islsm.16-OR-07. PMID 27721561
- [Background] Oh-hama T, Santander PJ, Stolowich NJ, Scott AI. Bacteriochlorophyll c formation via the C5 pathway of 5-aminolevulinic acid synthesis in Chloroflexus aurantiacus. FEBS Lett. 1991 Apr 9;281(1-2):173-6. doi: 10.1016/0014-5793(91)80386-h. PMID 2015889
- [Background] Ferraresi C, Huang YY, Hamblin MR. Photobiomodulation in human muscle tissue: an advantage in sports performance? J Biophotonics. 2016 Dec;9(11-12):1273-1299. doi: 10.1002/jbio.201600176. Epub 2016 Nov 22. PMID 27874264
- [Background] Alayat MS, Mohamed AA, Helal OF, Khaled OA. Efficacy of high-intensity laser therapy in the treatment of chronic neck pain: a randomized double-blind placebo-control trial. Lasers Med Sci. 2016 May;31(4):687-94. doi: 10.1007/s10103-016-1910-2. Epub 2016 Feb 25. PMID 26914684
- [Background] Stiglic-Rogoznica N, Stamenkovic D, Frlan-Vrgoc L, Avancini-Dobrovic V, Vrbanic TS. Analgesic effect of high intensity laser therapy in knee osteoarthritis. Coll Antropol. 2011 Sep;35 Suppl 2:183-5. PMID 22220431
- [Background] Karu T. Mitochondrial mechanisms of photobiomodulation in context of new data about multiple roles of ATP. Photomed Laser Surg. 2010 Apr;28(2):159-60. doi: 10.1089/pho.2010.2789. No abstract available. PMID 20374017
- [Background] Espejo-Antunez L, Tejeda JF, Albornoz-Cabello M, Rodriguez-Mansilla J, de la Cruz-Torres B, Ribeiro F, Silva AG. Dry needling in the management of myofascial trigger points: A systematic review of randomized controlled trials. Complement Ther Med. 2017 Aug;33:46-57. doi: 10.1016/j.ctim.2017.06.003. Epub 2017 Jun 15. PMID 28735825
- [Background] Segura-Perez M, Hernandez-Criado MT, Calvo-Lobo C, Vega-Piris L, Fernandez-Martin R, Rodriguez-Sanz D. A Multimodal Approach for Myofascial Pain Syndrome: A Prospective Study. J Manipulative Physiol Ther. 2017 Jul-Aug;40(6):397-403. doi: 10.1016/j.jmpt.2017.06.001. Epub 2017 Jul 21. PMID 28739020
- [Background] Desai MJ, Saini V, Saini S. Myofascial pain syndrome: a treatment review. Pain Ther. 2013 Jun;2(1):21-36. doi: 10.1007/s40122-013-0006-y. Epub 2013 Feb 12. PMID 25135034
- [Background] Borg-Stein J, Iaccarino MA. Myofascial pain syndrome treatments. Phys Med Rehabil Clin N Am. 2014 May;25(2):357-74. doi: 10.1016/j.pmr.2014.01.012. Epub 2014 Mar 17. PMID 24787338
- [Background] Xia P, Wang X, Lin Q, Cheng K, Li X. Effectiveness of ultrasound therapy for myofascial pain syndrome: a systematic review and meta-analysis. J Pain Res. 2017 Mar 7;10:545-555. doi: 10.2147/JPR.S131482. eCollection 2017. PMID 28331357
- [Background] Rodriguez-Perea A, Chirosa Rios LJ, Martinez-Garcia D, Ulloa-Diaz D, Guede Rojas F, Jerez-Mayorga D, Chirosa Rios IJ. Reliability of isometric and isokinetic trunk flexor strength using a functional electromechanical dynamometer. PeerJ. 2019 Oct 18;7:e7883. doi: 10.7717/peerj.7883. eCollection 2019. PMID 31695965
- [Background] Jerez-Mayorga D, Chirosa Rios LJ, Reyes A, Delgado-Floody P, Machado Payer R, Guisado Requena IM. Muscle quality index and isometric strength in older adults with hip osteoarthritis. PeerJ. 2019 Aug 7;7:e7471. doi: 10.7717/peerj.7471. eCollection 2019. PMID 31410316
- [Background] Knapstad MK, Nordahl SHG, Naterstad IF, Ask T, Skouen JS, Goplen FK. Measuring pressure pain threshold in the cervical region of dizzy patients-The reliability of a pressure algometer. Physiother Res Int. 2018 Oct;23(4):e1736. doi: 10.1002/pri.1736. Epub 2018 Aug 7. PMID 30088327
- [Background] Hanney WJ, Puentedura EJ, Kolber MJ, Liu X, Pabian PS, Cheatham SW. The immediate effects of manual stretching and cervicothoracic junction manipulation on cervical range of motion and upper trapezius pressure pain thresholds. J Back Musculoskelet Rehabil. 2017 Sep 22;30(5):1005-1013. doi: 10.3233/BMR-169573. PMID 28505955
- [Background] Lee B, Lee J, Yang J, Heo K, Hwang H, Kim B, Han D. The effects of stretching exercise for upper trapezius on the asymmetric rate of bite force. J Phys Ther Sci. 2015 Jul;27(7):2159-62. doi: 10.1589/jpts.27.2159. Epub 2015 Jul 22. PMID 26311945
- [Background] Palacios-Cena M, Wang K, Castaldo M, Guerrero-Peral A, Caminero AB, Fernandez-de-Las-Penas C, Arendt-Nielsen L. Assessment of deep dynamic mechanical sensitivity in individuals with tension-type headache: The dynamic pressure algometry. Eur J Pain. 2017 Sep;21(8):1451-1460. doi: 10.1002/ejp.1065. Epub 2017 Jun 2. PMID 28573720